CLINICAL TRIAL: NCT00334516
Title: Cortical Function in Primary Lateral Sclerosis and Amyotrophic Lateral Sclerosis
Brief Title: Brain Function in Primary Lateral Sclerosis and Amyotrophic Lateral Sclerosis
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060174; 06-N-0174
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2019-05-31 (Actual); Status verified 2015-08-03

CONDITIONS: Cerebral Cortex Dysfunction
Keywords: Motor Neuron Disease; Cognitive Testing; Movement-Related Potential; MRI; Neuropsychologic Testing; Primary Lateral Sclerosis; PLS; Amyotrophic Lateral Sclerosis; ALS; Healthy Volunteer; HV
MeSH Terms: conditions — Motor Neuron Disease; Amyotrophic Lateral Sclerosis

SUMMARY:
This study will test whether primary lateral sclerosis (PLS) and amyotrophic lateral sclerosis (ALS) affect parts of the brain responsible for thinking, planning, memory and emotion.

Healthy volunteers 18 years of age and older and patients with PLS and ALS may be eligible for this study.

Participants undergo the following procedures:

* Rating motor function: Subjects are asked to contract certain muscles in the face, arms and legs, to tap their finger on a keyboard rapidly, to walk 20 feet, and to read a paragraph out loud.
* Electroencephalography (EEG): The electrical activity of the brain (brain waves) is recorded while subjects tap their finger very slowly. For this test, electrodes are placed on the scalp using a cap or an adhesive substance. A conductive gel is used to fill the space between the electrodes and the scalp to ensure good contact.
* Surface electromyography (EMG): The electrical activity of the muscles is measured. Electrodes filled with a conductive gel are taped to the skin over the muscle tested.
* Neuropsychological testing: Testing may include questionnaires, pen-and-paper or computerized tests, and motor tasks.
* Magnetic resonance imaging (MRI): MRI uses a strong magnetic field and radio waves to produce images of the brain. The subject lies on a table that slides into the scanner. Scanning time varies from 20 minutes to 3 hours, with most scans lasting 45-90 minutes.

DETAILED DESCRIPTION:
Objective:

The goal of this study is to see whether patterns of cerebral cortex dysfunction differ in Primary lateral sclerosis (PLS) and amyotrophic lateral sclerosis (ALS). The function of several regions of the cerebral cortex will be assessed by clinical, physiological, and neuropsychological tests. Magnetic resonance imaging will be carried out in a subset of patients to explore the correlation between functional and anatomical measures of these cortical areas.

Study Population:

30 patients with Primary lateral sclerosis who meet the diagnostic criteria for PLS proposed by Pringle and 30 patients with ALS who fulfill the revised El Escorial criteria for probable or definite ALS.

30 healthy volunteers will be studied to provide training and practice in using the rating scales and to provide age-matched controls for EEG and imaging studies.

Design:

A screening examination will be carried out under protocol 01-N-0145 to determine eligibility. Patients and caregivers will return for two or three visits for sessions of neuropsychological testing, a structured clinical neuropsychiatric evaluation, ratings of motor and clinical function, and measurement of movement-related cortical potentials with EEG. A subset of patients will undergo MRI scans for quantitative anatomical measures of cortical regions.

Outcome Measures:

The primary outcome will be the classification of patients as normal or abnormal on neuropsychological testing of frontal cortex function. Correlations of the primary outcome with other variables - clinical measures of motor function, neuropsychiatric assessment will be examined. EEG measures of movement related cortical potentials and MR imaging findings will be analyzed in an exploratory fashion to determine whether these measures differ between PLS and ALS patients.

ELIGIBILITY:
* PRIMARY LATERAL SCLEROSIS INCLUSION CRITERIA:

Patients with PLS, aged 18 and older, must meet the diagnostic criteria proposed by Pringle (1992), incorporating Santa Clara (2004) consensus for pure PLS.

Clinical:

* Insidious onset in adulthood, progressive course
* No family history
* Disease duration greater than 3 years without lower motor neuron clinical signs
* Clinical signs restricted to corticospinal/corticobulbar tract dysfunction

Imaging:

* Brain MRI normal (except cortical atrophy)
* Normal cervical spine
* Negative chest X-ray, negative mammograms in women

EMG after 3 years, but within last 3 years, showing no active denervation.

Normal serological studies for serum chemistry, Vitamin B12, Vitamin E levels, very long-chain fatty acids.

Negative serology for syphilis, Lyme disease, HTLV 1 and 2.

AMYOTROPHIC LATERAL SCLEROSIS INCLUSION CRITERIA:

Patients with ALS, aged 18 and older, must fulfill the revised El Escorial criteria for probable or definite ALS.

* Probable ALS: Upper and Lower motor neuron signs are present in more than two regions, but some UMN signs must be rostral to LMN signs.
* Definite ALS: Upper and Lower motor neuron signs are present in more than three regions.

HEALTHY VOLUNTEERS INCLUSION CRITERIA:

Healthy adults, aged 18 and older, willing to participate, and able to give informed consent.

EXCLUSION CRITERIA:

Cognitive impairment of such severity that patients cannot provide assent to participate in the protocol. During the screening examination, we will question the patients to see if they understand that they are being evaluated, the types of tests we are using, and the response required. If they are unable to answer these questions, they will be excluded from the study.

History or evidence of co-existence of a second neurological disorder, such as stroke, epilepsy, Parkinson's disease, polio, ataxia or neuropathy.

History of traumatic brain injury, skull defects or neurosurgery.

Patients who fulfill the inclusion criteria for ALS and PLS but have the following conditions will be allowed to participate in cognitive studies and EEG studies, but will be excluded from MRI testing.

* Pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, or shrapnel fragments.
* Occupational exposure to metal fragments, as in welders and metal workers, which may lead to small fragments in the eye.
* Pregnancy. Women of childbearing potential will undergo urine pregnancy testing before MRI scanning.
* Fear of confined spaces.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2006-06-06; Study Completion 2015-08-03

CONTACTS AND LOCATIONS:
Overall Officials: Mary Kay Floeter, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Pringle CE, Hudson AJ, Munoz DG, Kiernan JA, Brown WF, Ebers GC. Primary lateral sclerosis. Clinical features, neuropathology and diagnostic criteria. Brain. 1992 Apr;115 ( Pt 2):495-520. doi: 10.1093/brain/115.2.495. PMID 1606479
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847
- [Background] Younger DS, Chou S, Hays AP, Lange DJ, Emerson R, Brin M, Thompson H Jr, Rowland LP. Primary lateral sclerosis. A clinical diagnosis reemerges. Arch Neurol. 1988 Dec;45(12):1304-7. doi: 10.1001/archneur.1988.00520360022005. PMID 3196189
- [Derived] Kwan JY, Jeong SY, Van Gelderen P, Deng HX, Quezado MM, Danielian LE, Butman JA, Chen L, Bayat E, Russell J, Siddique T, Duyn JH, Rouault TA, Floeter MK. Iron accumulation in deep cortical layers accounts for MRI signal abnormalities in ALS: correlating 7 tesla MRI and pathology. PLoS One. 2012;7(4):e35241. doi: 10.1371/journal.pone.0035241. Epub 2012 Apr 17. PMID 22529995
- [Derived] Iwata NK, Kwan JY, Danielian LE, Butman JA, Tovar-Moll F, Bayat E, Floeter MK. White matter alterations differ in primary lateral sclerosis and amyotrophic lateral sclerosis. Brain. 2011 Sep;134(Pt 9):2642-55. doi: 10.1093/brain/awr178. Epub 2011 Jul 28. PMID 21798965